CLINICAL TRIAL: NCT03229057
Title: Comparing the Effects of Oral Contraceptive Pills Versus Metformin in the Medical Management of Overweight/Obese Women With Polycystic Ovary Syndrome
Brief Title: Comparing the Effects of Oral Contraceptive Pills Versus Metformin
Acronym: COMET-PCOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anuja Dokras (Other)
Collaborators: Milton S. Hershey Medical Center (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Anuja Dokras, Professor of Obstetrics and Gynecology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 827819; 5R01HD091350-05 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-25 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: PCOS
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This will be a three-arm, double-blind, double-dummy, multicenter, prospective, randomized clinical trial comparing OCP vs. Metformin vs. OCP + Metformin on the prevalence of MetS in women with PCOS. This 6-month study will consist of a screening visit, followed by 6 study visits. No longer term follow-up is planned.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- OCP + Placebo (Active Comparator): The OCP will be started on the first Sunday after spontaneous or induced menses. All subjects with no menses the 4 weeks before randomization will be given medroxyprogesterone acetate after a negative pregnancy test (in order to induce menses). Placebo pills will be administered to individuals randomized to OCP only in order to maintain study blinding.
  Interventions: Drug: OCP + Placebo
- Metformin + Placebo (Active Comparator): Metformin will be initiated in a step-up fashion on cycle day 1-3 of spontaneously or induced menses. Extended release pills will be utilized as they are associated with fewer gastrointestinal side effects. Subjects will begin with one tablet of metformin every night for 5 days, eventually building up to 4 tablets every night, with the maximum dose of metformin being 2000 mg. Placebo pills will be administered to individuals randomized to metformin only in order to maintain study blinding.
  Interventions: Drug: Metformin + Placebo
- OCP + Metformin (Experimental): The OCP will be started on the first Sunday after spontaneous or induced menses. All subjects with no menses the 4 weeks before randomization will be given medroxyprogesterone acetate after a negative pregnancy test (in order to induce menses). Metformin will be initiated in a step-up fashion on cycle day 1-3 of spontaneously or induced menses. Extended release pills will be utilized as they are associated with fewer gastrointestinal side effects. Subjects will begin with one tablet of metformin every night for 5 days, eventually building up to 4 tablets every night, with the maximum dose of metformin being 2000 mg.
  Interventions: Drug: OCP + Metformin

INTERVENTIONS:
Drug: OCP + Metformin — This will be a three-arm, double-blind, double-dummy, multicenter, prospective, randomized clinical trial comparing OCP vs. Metformin vs. OCP + Metformin on the prevalence of MetS in women with PCOS. This 6-month study will consist of a screening visit, followed by 6 study visits (Subjects will undergo 6 in person study visits and life style modification counseling regarding diet and exercise. Phone contact will be made 2 weeks after randomization and at the end of each month when there is no in person visit to ensure study compliance with medications, keeping study logs and to review side effects). No longer term follow-up is planned.
  Arms: OCP + Metformin
Drug: OCP + Placebo — This will be a three-arm, double-blind, double-dummy, multicenter, prospective, randomized clinical trial comparing OCP vs. Metformin vs. OCP + Metformin on the prevalence of MetS in women with PCOS. This 6-month study will consist of a screening visit, followed by 6 study visits (Subjects will undergo 6 in person study visits and life style modification counseling regarding diet and exercise. Phone contact will be made 2 weeks after randomization and at the end of each month when there is no in person visit to ensure study compliance with medications, keeping study logs and to review side effects). No longer term follow-up is planned.
  Arms: OCP + Placebo
Drug: Metformin + Placebo — This will be a three-arm, double-blind, double-dummy, multicenter, prospective, randomized clinical trial comparing OCP vs. Metformin vs. OCP + Metformin on the prevalence of MetS in women with PCOS. This 6-month study will consist of a screening visit, followed by 6 study visits (Subjects will undergo 6 in person study visits and life style modification counseling regarding diet and exercise. Phone contact will be made 2 weeks after randomization and at the end of each month when there is no in person visit to ensure study compliance with medications, keeping study logs and to review side effects). No longer term follow-up is planned.
  Arms: Metformin + Placebo

SUMMARY:
To determine the effect of Oral Contraceptive Pills (OCP) verses Metformin verses OCP and Metformin on the prevalence of Metabolic Syndrome (MetS) and its components in overweight/obese women with Polycystic Ovary Syndrome (PCOS).

The combination of OCP and metformin (OCP, through lowering androgens, and metformin, through improvement in insulin sensitivity) will affect the prevalence of MetS, thereby altering the risk profile for the development of diabetes and possible cardiovascular disease (CVD) in young women with PCOS.

DETAILED DESCRIPTION:
The intervention will consist of randomizing subjects to one of three arms. Subjects will either be assigned to OCP + Placebo, Metformin + Placebo or OCP + Metformin. Metformin will be initiated in a step-up fashion on cycle day 1-3 of spontaneously or induced menses. Extended release pills will be utilized as they are associated with fewer gastrointestinal side effects. Subjects will begin with one tablet of metformin every night for 5 days, eventually building up to 4 tablets every night, with the maximum dose of metformin being 2000 mg. In regards to OCP, previous randomized clinical trials (RCTs) have shown that 20mcg ethinyl estradiol/norethindrone 1.0 mg was well tolerated. The study will utilize a 20mcg OCP but a less androgenic third generation progestin (desogestrel 0.15mg) with potentially lesser impact on lipids and insulin sensitivity. The OCP will be started on the first Sunday after spontaneous or induced menses. All subjects with no menses the 4 weeks before randomization will be given medroxyprogesterone acetate after a negative pregnancy test (in order to induce menses). Placebo pills will be administered to individuals randomized to OCP or metformin only in order to maintain study blinding. Subjects will undergo 6 in person study visits and life style modification counseling regarding diet and exercise. Phone contact will be made 2 weeks after randomization and at the end of each month when there is no in person visit to ensure study compliance with medications, keeping study logs and to review side effects

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 to ≤ 40 years of age (at the time of screening), with hyperandrogenic PCOS.
2. Subjects will be diagnosed with PCOS defined by the most recent Rotterdam criteria based on:

   1. androgen excess (defined as an elevated serum T level or hirsutism, based on a Ferriman Gallwey score > 8 (note: > 2 for women of Asian descent)

      AND either:
   2. history of chronic anovulation (8 or fewer periods per year)

      AND/OR
   3. polycystic ovaries.
3. BMI ≥ 25 kg/m² to ≤ 48 kg/m² obtained at screening visit.
4. In good general health.
5. Willing to avoid pregnancy for the duration of the study.

Exclusion Criteria:

1. Current pregnancy or desire of pregnancy during course of study
2. Currently breastfeeding
3. Known 21 hydroxylase deficiency
4. Untreated thyroid disease (TSH <0.45 mlU/mL and > 4.5 mlU/mL)
5. Untreated hyperprolactinemia (2 Levels>30 ng/ml at least one week apart)
6. Type 1 or type 2 Diabetes Mellitus (elevated fasting serum glucose >126mg/dL on two occasions, poorly controlled diabetes (HgbA1C>6.5%), currently receiving anti-diabetic agents, or currently receiving metformin for treatment of diabetes
7. Liver disease (AST/ALT>2 times normal or a total bilirubin >2.5 mg/dL)
8. Renal disease (BUN>30 mg/dL or serum creatinine >1.4 mg/dL)
9. Anemia (hemoglobin <10 mg/dL)
10. History of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident
11. Current history of alcohol abuse (>14drinks/week)
12. Poorly controlled hypertension defined as average systolic blood pressure >= 150 mm Hg or average diastolic >=100 mm Hg obtained on three measurements obtained 5 minutes apart. If treated, average systolic blood pressure >=140 mm Hg or average diastolic >=90 mm Hg
13. Patients with a history of, or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma
14. TG>200mg/dl
15. Use of lipid lowering or weight loss agents (subjects may wash out from weight loss agents)
16. Current use of oral contraceptives, depo progestin, or hormonal implants
17. Participation in any study of an investigational drug or device or biological agent within 30 days
18. Suspected adrenal or ovarian tumor secreting androgens
19. Suspected Cushing's syndrome
20. Bariatric surgery procedure in the recent past (<12 months)
21. Absolute contraindications to the use of hormonal contraceptives or metformin,

23. Subjects who are unable to comply with the study procedures, for instance due to mental illness, substance abuse, or participation in other studies.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Dokras, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Penn State/ Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dokras A, Coutifaris C, Remaley AT, Mehta NN, Playford MP, Kunselman AR, Stetter CC, Dodson WC, Legro RS. Impact of combined hormonal contraceptives and metformin on metabolic syndrome in women with hyperandrogenic polycystic ovary syndrome and obesity: The COMET-PCOS randomized clinical trial. PLoS Med. 2025 Dec 8;22(12):e1004662. doi: 10.1371/journal.pmed.1004662. eCollection 2025 Dec. PMID 41359669
- See also: Related Info — http://pennhealth.com/fertility/
- See also: Related Info — http://whcrc.upenn.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Started | 79 | 81 | 80
End of study outcome | 59 | 65 | 63
Completed | 52 | 60 | 57
Not Completed | 27 | 21 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin | Total
Number analyzed (Participants) | 79 | 81 | 80 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (4.8) | 30.1 (5.3) | 29.2 (5.4) | 29.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 81 | 80 | 240
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 17 | 14 | 42
  Not Hispanic or Latino | 68 | 64 | 66 | 198
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 19 | 16 | 19 | 54
  White | 53 | 59 | 57 | 169
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Menses per year [Mean (Standard Deviation); unit: menses per year] — Population: Baseline menses data were missing for 7 participants.
  menses per year
    number analyzed (Participants) | 75 | 79 | 79 | 233
    (all) | 4.7 (3.2) | 5.7 (3.8) | 4.8 (3.3) | 5.1 (3.4)
Percentage of Nulliparous [Count of Participants; unit: Participants] | 56 | 57 | 58 | 171
Count of Current Smokers [Count of Participants; unit: Participants] | 6 | 5 | 5 | 16
Percentage of Participants on Hypertension Medications [Count of Participants; unit: Participants] | 7 | 2 | 2 | 11
Percentage of Participants with Prediabetes, based on HbA1C [Count of Participants; unit: Participants] | 27 | 27 | 27 | 81
Waist measurement [Mean (Standard Deviation); unit: cm] | 108.0 (12.8) | 107.4 (15.6) | 109.0 (16.4) | 108 (15.0)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 116.8 (9.8) | 116.9 (10.1) | 117.0 (8.4) | 116.9 (9.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHG] | 76.8 (7.3) | 77.7 (6.4) | 76.9 (6.3) | 77.1 (6.8)
Fasting glucose value from safety labs [Mean (Standard Deviation); unit: mg/dL] | 78.1 (14.7) | 77.6 (17.0) | 74.2 (15.8) | 76.6 (15.9)
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 102.0 [75.0 to 137.0] | 90.0 [66.0 to 121.0] | 97.0 [68.5 to 152.0] | 97.5 [69.0 to 137.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Metabolic Syndrome After 6 Months of Treatment Metformin or OCP+Metformin for 6 Months.
Description: Our primary goal is to determine the effect of 6 months' treatment with OCP vs. metformin vs. OCP + metformin on prevalence of MetS and its components in overweight / obese women. Implicit in the primary aim is clearly defining MetS, by NCEP ATPIII criteria as the presence of at least 3 of the following 5 criteria: TG≥150mg/dl, HDL-C<50mg/dl, BP≥130/≥85mmHg, WC>88cm and fasting glucose≥100mg/dl; and the goal of tracking safety of our interventions at all Phases of the study (through safety lab evaluations, vital signs and diaries)
Time Frame: Baseline and 6 months
Population: Includes all participants who completed an end of study visit greater than or equal to 16 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 59 | 65 | 63
Participants | 17 | 17 | 18

2. Secondary Outcome: Changes in Serum Apoliprotein B From Baseline to 6 Months
Description: This will be measured by NMR spectroscopy
Time Frame: Baseline and 6 months
Population: Uses all available data, Intent to Treat
Measure: Mean (Inter-Quartile Range); unit: g/L
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
g/L | .03 [-0.02 to 0.06] | 0.003 [-0.03 to 0.04] | 0.05 [0.01 to 0.09]

3. Secondary Outcome: Changes in Serum Adipokines in the 3 Arms
Description: Serum adipokines to be measured are adiponectin and leptin. These changes will be correlated with changes in serum and androgens and markers of insulin sensitivity.
Time Frame: Baseline and 6 months
Population: The study team planned to complete this outcome, however, we did not have funding to complete the outcome and there is no plan to run this analysis in the future. Therefore we have no results to report, nor will we in the future.
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Changes in Total Body Fat Distribution in the 3 Arms From Baseline to 6 Months
Description: Body fat distribution will be measured by DXA. These changes will be correlated with changes in serum and androgens and markers of insulin sensitivity
Time Frame: Baseline and 6 months
Population: Uses all available data, Intent to Treat
Measure: Mean (Inter-Quartile Range); unit: kg
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
kg | -0.83 [-1.65 to -0.01] | -0.48 [-1.24 to 0.28] | 0.06 [-0.70 to 0.82]

5. Secondary Outcome: Changes in Total Triglyceride-Rich Lipoprotein (TRLP) From Baseline to 6 Months
Description: This will be measured by NMR spectroscopy
Time Frame: Baseline and 6 months
Measure: Mean (Inter-Quartile Range); unit: mol/L
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
mol/L | -2.26 [-0.02 to 0.06] | 6.33 [-5.35 to 18.02] | 10.24 [-1.70 to 22.18]

6. Secondary Outcome: Changes in Serum Marker of Inflammation: Free Fatty Acids.
Description: Measured by change in Free Fatty Acids
Time Frame: Baseline and 6 months
Population: Uses all available data, Intent to Treat
Measure: Mean (Inter-Quartile Range); unit: mEq/L
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
mEq/L | 0.04 [-0.02 to 0.10] | -0.03 [-0.09 to 0.03] | 0.09 [0.03 to 0.15]

7. Secondary Outcome: Changes in Quality of Life Parameters for Body Hair in All 3 Arms as Assessed by PCOSQ From Baseline to 6 Months
Description: QOL will be measured by the Polycystic Ovary Syndrome Questionnaire (PCOSQ) Body Hair domain which has 5 items rated on a 7 point likert scale with a lower score representing a decreased quality of life. The total range is 7 to 35.
Time Frame: Baseline and 6 months
Population: Uses all available data, Intent to Treat
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
score on a scale | 0.74 [0.46 to 1.02] | 0.26 [-0.01 to 0.53] | 0.62 [0.35 to 0.90]

8. Secondary Outcome: Changes in Visceral Body Fat Distribution in the 3 Arms
Description: as for outcome 4
Time Frame: Baseline and 6 months
Population: Uses all available data, Intent to Treat
Measure: Mean (Inter-Quartile Range); unit: g
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
g | -167 [-264 to -71] | -86 [-176 to 4] | -58 [-148 to 32]

9. Secondary Outcome: Changes in Quality of Life Parameters for Weight in All 3 Arms as Assessed by PCOSQ From Baseline to 6 Months
Description: QOL will be measured by the Polycystic Ovary Syndrome Questionnaire (PCOSQ) Weight domain which has 5 items rated on a 7 point likert scale with a lower score representing a decreased quality of life. The total range is 7 to 35.
Time Frame: Baseline and 6 months
Population: Uses all available data, Intent to Treat
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 79 | 81 | 80
score on a scale | 0.72 [0.37 to 1.07] | 0.34 [0.01 to 0.68] | 0.62 [0.35 to 0.90]

10. Secondary Outcome: Change in HDL-C Function
Description: This will be assessed by measuring reverse cholesterol efflux capacity using validated ex vivo system.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected for 7 months.
Arm/Group | OCP + Placebo | Metformin + Placebo | OCP + Metformin
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/81 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/79 | 3/81 | 3/80
Other Adverse Events (participants affected / at risk) | 71/79 | 76/81 | 78/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCP + Placebo (N=79) | Metformin + Placebo (N=81) | OCP + Metformin (N=80)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Gastroenteritis resulting in dehydration
Surgical Intervention (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Exploratory laparoscopy for severe lower abdominal pain
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Hospitalization for sever depression
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Pregnancy with miscarriage at 20 weeks, 5 days
Hospitalization (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — Ongoing bleeding despite medical management. Admitted for blood transfusion and D&C.
Hospitalization (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Gall bladder attack with surgery
Medical intervention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Headache/vision problems diagnosed to be idiopathic intracranial hypertension
Hospitalization (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Cholecystectomy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCP + Placebo (N=79) | Metformin + Placebo (N=81) | OCP + Metformin (N=80)
Diarrhea (Gastrointestinal disorders) | 27 (31) | 52 (78) | 52 (67)
Nausea (Gastrointestinal disorders) | 29 (31) | 34 (42) | 37 (44)
Abdominal Pain/Cramping (Gastrointestinal disorders) | 10 (11) | 27 (30) | 20 (22)
Vomiting (Gastrointestinal disorders) | 8 (8) | 20 (21) | 18 (21)
Abdominal Bloating (Gastrointestinal disorders) | 10 (11) | 9 (10) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 5 (7) | 12 (12)
Decreased Appetite (Gastrointestinal disorders) | 3 (3) | 3 (4) | 7 (7)
Flatulence (Gastrointestinal disorders) | 6 (6) | 9 (9) | 4 (4)
Vaginal Bleeding/Spotting (Reproductive system and breast disorders) | 19 (22) | 2 (3) | 7 (8)
Dysmenorrhea (Reproductive system and breast disorders) | 15 (21) | 9 (14) | 11 (12)
Breast Symptoms (Reproductive system and breast disorders) | 7 (9) | 2 (2) | 5 (8) — Breast tenderness/pain/swelling
Dizziness (Nervous system disorders) | 3 (3) | 6 (8) | 4 (4)
Headache/Migraine (Nervous system disorders) | 21 (44) | 21 (34) | 21 (27)
Mood Swings/Depression (Psychiatric disorders) | 10 (11) | 3 (3) | 3 (3)
Joint/muscle pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 16 (16) | 14 (16) | 8 (8)
COVID infection/symptoms after exposure (Infections and infestations) | 7 (7) | 3 (3) | 4 (4)
Fatigue (General disorders) | 4 (4) | 9 (9) | 6 (6)

LIMITATIONS AND CAVEATS:
Two outcomes, Changes in HDL-C function assessed by measuring reverse cholesterol efflux capacity using validated ex vivo system and serum adipokines which are to be measured are adiponectin and leptin. We are currently looking for a vendor to run these assays.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT03229057/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03229057/ICF_002.pdf